CLINICAL TRIAL: NCT05252715
Title: A Single-center, Randomized, Blind, Positive Control Phase III Clinical Trial to Evaluate Immunogenicity and Safety of Meningococcal ACYW135 Polysaccharide Conjugate Vaccine in Healthy Volunteers Aged From 3 to 5 Months
Brief Title: Immunogenicity and Safety of Meningococcal ACYW135 Polysaccharide Conjugate Vaccine in Volunteers Aged From 3 to 5 Months
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020040C-1
Record Dates: First submitted 2022-02-13; First posted 2022-02-23 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Meningitis, Meningococcal
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meningococcal ACYW135 Polysaccharide Conjugate Vaccine (Experimental): Meningococcal ACYW135 Polysaccharide Conjugate Vaccine, 20 µg/dose. Primary vaccination at 0, 1 and 2 months of age, respectively. Booster vaccination at 18 months of age.
  Interventions: Biological: Meningococcal ACYW135 Polysaccharide Conjugate Vaccine
- Meningococcal A and C Polysaccharide Conjugate Vaccine (Active Comparator): Meningococcal A and C Polysaccharide Conjugate Vaccine, 20 µg/dose. Primary vaccination at 0, 1 and 2 months of age, respectively.
  Interventions: Biological: Meningococcal A and C Polysaccharide Conjugate Vaccine

INTERVENTIONS:
Biological: Meningococcal ACYW135 Polysaccharide Conjugate Vaccine — Single intramuscular dose contains 5 µg each of Serogroup A, C, Y, and W135 meningococcal polysaccharide combined with tetanus toxoid.
  Arms: Meningococcal ACYW135 Polysaccharide Conjugate Vaccine
Biological: Meningococcal A and C Polysaccharide Conjugate Vaccine — Single intramuscular dose contains 10 µg each of Serogroup A and C meningococcal polysaccharide combined with tetanus toxoid.
  Arms: Meningococcal A and C Polysaccharide Conjugate Vaccine

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of Meningococcal ACYW135 Polysaccharide Conjugate Vaccine in healthy volunteers aged from 3 to 5 months.

ELIGIBILITY:
Inclusion Criteria:

For primary vaccination

* Subjects aged 3-5 months;
* Subjects should be full-term (37-42 weeks of gestation) and their birth weight should meet the requirements (2500g ≤ body weight ≤ 4000g);
* Axillary body temperature ≤ 37.0 ℃;
* The guardian signs the informed consent form;
* The guardian and his family agree to comply with the requirements of the clinical trial protocol;
* Subjects who have not been vaccinated with meningococcal group A and C conjugate vaccine at the aged of 3-5 months;
* Subjects who had no history of other live vaccines within 14 days before vaccination and no history of other inactivated vaccines within 7 days;

For booster vaccination

* Infants in the experimental group who have completed primary immunization in this clinical trial and reach the age of 18 months;
* The guardian and his family agree to comply with the requirements of the clinical trial protocol.

Exclusion Criteria:

For primary vaccination

* Test-tube baby who is suffering from perianal abscess, severe eczema or pathological jaundice;
* History of severe allergic reactions requiring medical intervention (such as swelling of mouth and throat, dyspnea, hypotension or shock);
* A clearly diagnosed history of thrombocytopenia or other coagulation disorders that may cause contraindications to intramuscular injection;
* History of Abnormal production process, asphyxia rescue, or congenital malformation, serious developmental disorder, serious genetic defect, serious malnutrition or serious chronic disease;
* Have been diagnosed as infectious diseases, such as tuberculosis, viral hepatitis or their parents infected with human immunodeficiency virus (HIV);
* Have progressive nervous system diseases such as encephalopathy, epilepsy, convulsions or related family history;
* History of acute disease, severe chronic disease, acute attack of chronic disease and fever (axillary body temperature ≥ 38.0 ℃) or take antipyretic, analgesic and antiallergic drugs (such as acetaminophen, ibuprofen, aspirin, etc.) in the past 3 days;
* History of using illegal drugs (receiving systemic corticosteroid treatment≥2mg/kg/day through any route of administration, and using ≥14 days, such as prednisone, inhaled hormone budesonide, fluticasone, etc., or receiving other immunosuppressants, such as cyclophosphamide, etc.);
* History of using immunoglobulins and / or any blood products (except hepatitis B immunoglobulin) within 3 months before enrollment;
* Plan to participate or be participating in any other drug clinical research;
* According to the judgment of the investigator, the subject has any other factors that are not suitable for participating in the clinical trial.

For booster vaccination

* The subjects were vaccinated with any meningococcal vaccine after primary immunization and before blood collection of booster immunization;
* The subjects have been known or suspected to have immunological defects since participating in this clinical trial, including being treated with immunosuppressants (such as chemotherapy, corticosteroids, antimetabolics, cytotoxic drugs, etc.) and HIV infection;
* History of using immunoglobulins and / or any blood products (except hepatitis B immunoglobulin) within 3 months before booster immunization;
* According to the judgment of the investigator, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 3 Months to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2021-12-18 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2024-09-18 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity study of Meningococcal ACYW135 Polysaccharide Conjugate Vaccine as assessed by positive conversion rate | 30 day after each vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Lin Du, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (2):
- China (2):
  - Liujiang Center for Disease Control and Prevention, Liuchow, Guangxi
  - Binyang Center for Disease Control and Prevention, Nanning, Guangxi